CLINICAL TRIAL: NCT06764797
Title: Investigating the Efficacy of Combining Virtual Reality-Based Mirror Therapy and Transcranial Direct Current Stimulation to Improve Upper Limb Recovery in Patients with Stroke
Brief Title: Investigating the Efficacy of Combining Virtual Reality-Based Mirror Therapy (VRMT) and Transcranial Direct Current Stimulation (tDCS) to Improve Upper Limb Recovery in Patients with Stroke
Acronym: tDCS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: King Fahad Medical City (Other Government); King Saud Medical City (Other Government)
Responsible Party: Principal Investigator, Dr. Alaa Albishi, Associate professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-23-7496; Not funded (Other: Not funded)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Stroke Rehabilitaion; Stroke
Keywords: Virtual reality, Mirror therapy, non invasive brain stimulation, tDCS, stroke; transcranial direct current stimulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- anodal tDCS combined with VRMT (Experimental): 20 minutes of anodal tDCS combined with 45 minutes of VRMT
  Interventions: Device: Transcranial Direct Current Stimulation compined with virtual reality based mirror therapy
- Anodal tDCS alone (Active Comparator): 20 minutes of anodal tDCS alone
  Interventions: Device: Transcranial Direct Current Stimulation
- VRMT alone, Sham tDCS (Active Comparator): 45 minutes of VRMT alone, For the sham-tDCS, the current flow will be terminated after 30 seconds.
  Interventions: Device: Virtual reality
- Conventional Physical therapy alone, Sham tDCS (Sham Comparator): 45 minutes of conventional physical therapy, For the sham-tDCS, the current flow will be terminated after 30 seconds.
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — tDCS will be used during the sessions. The anodal tDCS (2 mA) will be applied for 20 minutes. Continuous, direct currents. The anodal electrode will be positioned over the ipsilesional primary motor cortex (M1) (C3 or C4, international 10-20 system) of the affected hemisphere and the cathodal electrode over the contralateral orbit.
  Arms: Anodal tDCS alone
Device: Virtual reality — The VRMT group will receive VRMT game-based training using their non-affected upper limb. using a semi-immersive motion-tracking device.
  Arms: VRMT alone, Sham tDCS
Device: Transcranial Direct Current Stimulation compined with virtual reality based mirror therapy — 20 minutes of tDCS during 45 minutes of VRMT games.
  Arms: anodal tDCS combined with VRMT
Other: Conventional physical therapy — 45 minutes of conventional physical therapy with sham tDCS
  Arms: Conventional Physical therapy alone, Sham tDCS

SUMMARY:
This study will investigate whether combining virtual reality-based mirror therapy (VRMT) and transcranial direct current stimulation (tDCS) alongside conventional physical therapy (CPT) will significantly improve hand function for patients with stroke compared to using VRMT or tDCS alone.

DETAILED DESCRIPTION:
More than half of stroke survivors suffer from upper-limb dysfunction that persists years after stroke, negatively impacting patients' independence and, therefore, affecting their quality of life. Motor rehabilitation is required after a stroke to facilitate motor recovery. More importantly, finding new ways to maximize patients' motor recovery is a core goal of stroke rehabilitation. Thus, researchers have explored the potential benefits of using advanced technologies such as virtual reality-based mirror therapy (VRMT) and transcranial direct current stimulation (tDCS) to boost the brain's responses to interventions and maximize the effects of rehabilitation to improve upper-limb recovery post-stroke. However, the potential impact of combining VRMT and tDCS on upper limb functions for patients with stroke has not been explored. Therefore, the goal of this study is to investigate whether combining virtual reality-based mirror therapy (VRMT) with transcranial direct current stimulation (tDCS) alongside conventional physical therapy (CPT) will significantly improve hand function for patients with stroke compared to using VRMT or tDCS alone.

The participants will be randomly assigned into one of the four groups: (1) the anodal tDCS + VRMT group, (2) the anodal tDCS alone group, (3) the VRMT alone with sham tDCS group, and (4) the CPT with sham tDCS group. All groups will receive CPT as part of the treatment. Functional scales will be used before and after the intervention to assess upper motor functions. These measures include the Fugl-Meyer Assessment, Wolf Motor Function Test, Box and Block Test, Nine-Hole Pegboard Test, and Stroke Impact Scale-16 (SIS-16). In addition, physiological measures such as transcranial magnetic stimulation (TMS) and task-based fMRI.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Stroke patients with unilateral cerebral infarction or hemorrhage, more than three months following the stroke.
* Adequate cognitive ability to follow instructions (The Arabic version of the Mini-Mental State Examination scores > 24).
* Modified Ashworth scale score < 3.
* Fugl-Meyer Assessment (FMA) score of 10-58 indicating moderate-to-severe arm impairment.

Exclusion Criteria:

* visual impairment and field defect or hemi-sensory inattention and unilateral neglect.
* Wernicke's aphasia, or global aphasia, leads to difficulty following instructions.
* Any contraindication to NIBS.
* Other neurological conditions or participation in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-21 (Estimated)

PRIMARY OUTCOMES:
Fugl-Mayer Upper limb assessment (FMA) | at baseline, and after 2 weeks, and after intervention ( 4 weeks).
  FMA is a performance-based impairment measure particular to strokes, designed to assess motor functioning, balance, sensory, and joint functionality. It consists of five domains, which have 155 total items. The full potential scale score is 226. Scale items are scored based on the ability to finish the item using a 3-point ordinal scale. Motor score: from 0 to 100, 66 points for the upper extremity and 34 points for the lower extremities.
Wolf motor function test (WMT) | at baseline, and after 2 weeks, and after intervention ( 4 weeks).
  WMT, consisting of timed and practical tasks, measures the motor function of the upper extremity (UE). The WMFT has 17 items in the most common version. The first six items involved timed functional tasks; items 7 and 14 were strength tests, and the final nine analyzed the participants' movement quality while carrying out various tasks. Items scored on a 6-point scale, with lower scores indicating lower levels of functioning.
box and blocks test (BBT) | at baseline, and after 2 weeks, and after intervention ( 4 weeks).
  BBT assesses manual dexterity of the hand. It requires subjects to lift and release 2.5 cm³ cubes to move them from one compartment to another. BBT comprises 150 blocks. The test should begin with the unaffected upper limb to practice and record baseline values. The score is defined as the number of blocks transferred correctly within 60 seconds.
Nine-Hole Peg Test (NHPT) | at baseline, and after 2 weeks, and after intervention ( 4 weeks).
  NHPT was developed to assess finger dexterity. It is made up of a nine-peg square board. The board has holes on one end for the pegs to fit into, and it also has a shallow circular dish on the other for storing the pegs. The patient is instructed to quickly insert the pegs into the holes on the board after taking each one out of a container as part of the NHPT. Then, one by one, clients must bring the pegs out of the holes and put them back into the container. Scoring is according to how long it took them to finish the test activity, measured in seconds.

SECONDARY OUTCOMES:
Stroke impact scale-16 (SIS-16) | at baseline, and after 2 weeks, and after intervention ( 4 weeks).
  SIS is a self-report health status measure specific to the stroke population. It consists of 16 items from the four physical domains (strength, hand function ADL/IADL, and mobility).
transcranial magnetic stimulation (TMS) | at baseline, and after intervention ( 4 weeks).
  TMS measures cortical excitability, which is non-invasive magnetic stimulation using brief-duration, fast-pulsating, or pulsed magnetic fields to induce electrical currents targeted at spatially separate parts of the cerebral cortex using a computerized, electromechanical medical device.
Functional magnetic resonance imaging (fMRI) | at baseline, and after intervention ( 4 weeks).
  fMRI technique uses MRI technology to evaluate brain activity by looking for variations in blood flow. The coupling between cerebral blood flow and neuronal activation is the basis for this method. The participants will be trained on the task before the experimental session. A block design will be used in the fMRI scan; each fMRI scan lasts for 6 minutes, divided into six blocks with an interval of 30 seconds of task, 15 repeated contractions, each contraction lasting 2 seconds, interspersed with 30 seconds of rest.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M. Albishi, Doctor of Philosophy, Principal Investigator — King Saud University
Locations (2):
- Saudi Arabia (2):
  - King fahad medical city, Riyadh, Riyadh Region
  - King Khalid University Hospital, Riyadh, Riyadh Region